CLINICAL TRIAL: NCT05729334
Title: Clinical Investigation EUCLIDES-01 for the Calculation of the Area of Skin Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skilled Skin S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CIP-EUCLIDES-01
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Skin Lesion; Traumatic Ulcer; Hematoma; Pressure Ulcer; Venous Ulcer; Arterial Ulcer; Diabetic Neuropathic Ulcer; Ischemic Ulcer; Surgical Wound; Ulcer, Skin; Diabetic Foot Ulcer
Keywords: lesion skin; skin lesion; skin ulcer; wound area measurement; access; app; assessment; availability; correlation; mobile app; pressure ulcer; reliability; reproducibility; validity; wound; wound assessment; skin lesion area; measurement; calculation; Moisture Associated Skin Damage (MASD)
MeSH Terms: conditions — Hematoma; Pressure Ulcer; Varicose Ulcer; Surgical Wound; Skin Ulcer; Diabetic Foot; Alzheimer Disease; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects with skin lesions who meet all inclusion criteria and none of the exclusion criteria (Experimental): Subjects with skin lesions who meet all inclusion criteria and none of the exclusion criteria.
  Interventions: Device: Clinicgram Euclides

INTERVENTIONS:
Device: Clinicgram Euclides — Clinicgram Euclides is a software that allows automated calculation of the area of skin lesions using a mobile device. Three different photographs will be taken of the subject's skin lesion. The area of the skin lesion will be calculated using the photograph of the skin lesion, and:
  * for EUCLIDES 2D, an external marker. The investigator will outline the skin lesion and the external marker in the photograph prior to the calculation of the skin lesion area.
  * for EUCLIDES 3D, a two reference points selected by the investigator.

SUMMARY:
The aim of this clinical investigation is to collect skin lesion area data for the comparison of the agreement among the results obtained between the following three wound area measurement methods:

* Ruler using the Kundin method,
* Investigational software Clinicgram Euclides
* Digital planimetry with Adobe Photoshop

The clinical data retrieved in this study will allow the clinical validation of the safety and safety of the investigation software Clinicgram Euclides.

DETAILED DESCRIPTION:
The aim of the clinical investigation EUCLIDES-01 is to collect skin lesion area data for the comparison of the agreement among the results obtained between the following three skin lesion area measurement methods:

* Ruler using the Kundin method,
* Investigational software Clinicgram Euclides
* Digital planimetry with Adobe Photoshop

Clinicgram Euclides is a software that allows automatic calculation of skin lesion areas using a mobile device. It has two modes of operation (Euclides 2D and Euclides 3D).

The sample size is 65 subjects. Up to three skin lesions can be included from the same subject. For this reason, the number of subjects may be smaller if more than one skin lesion is measured in certain subjects.

EUCLIDES-01 is a pre-market, prospective, single-center, non-randomized clinical investigation with one arm of subjects intended to collect skin lesion area data for the comparison of the agreement among the results obtained between the three above-mentioned skin lesion area measurement methods.

No patient follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must give written informed consent prior to any procedure related to the clinical investigation.
2. Adult person 18 years of age or older.
3. The subject has an external skin lesion whose length and width can be measured with a 15-centimeter ruler.
4. The subject's external skin lesion can be measured with a perpendicular camera approach (90 degrees).
5. The subject has an external skin lesion located in an area that does not include an edge or curvature of the body, and that has no parts hidden by any device or treatment.
6. The subject has one or more isolated skin lesion(s) that allows for an individual capture and analysis process for each lesion.
7. Subjects are able to tolerate changes in position for at least 2 minutes in the area where the skin lesion is located.
8. Subjects can hold still, or not be prevented by pain from having still, for at least 10 seconds for the taking of the skin lesion photograph.

Exclusion Criteria:

1. The subject is currently participating in another clinical investigation.
2. Pregnant or breastfeeding women. Subjects who have medical, social, or psychological conditions that, in the opinion of the investigator, could limit the subject's ability to participate in the investigation or impact the scientific robustness of the clinical investigation results.

4. Subjects who have neoplastic, tumor, or pre-cancerous skin lesions. 5. Subjects presenting skin carcinomas or other skin lesions of confirmed malignancy (after differential diagnosis and screening of the potentially malignant lesion by clinical gross dermatology, dermatoscopy, microscopic dermatopathology, biopsy, or similar).

6. Subjects presenting skin lesions with excessive exudate that may obscure part of the skin lesion and its outline.

7. Subjects who suffer from movement disorders in the area where the skin lesion is located.

8. Subjects who may have allergies to the plastic of the external caliper or other skin irritations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2023-02-12 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Agreement of the skin lesion area measurements between two methods of routine clinical practice and the investigational software Clinicgram Euclides. | 1 day
  To assess the agreement/concordance of skin lesion area measurements between:
  * the investigational software Clinicgram Euclides and digital planimetry using Adobe Photoshop, and
  * the investigational software Clinicgram Euclides and the ruler measurement using the Kundin method.
Reproducibility of Clinicgram Euclides in the automatic calculation of skin lesion areas using different mobile devices. | 1 day
  To assess the reproducibility of Clinicgram Euclides in the e of skin lesion area measurements using two different mobile devices: an iPhone and an iPad.
Repeatability of Clinicgram Euclides in the automatic calculation of skin lesion areas between two measurements performed by the same investigator. | 1 day
  To assess the repeatability of Clinicgram Euclides in the automatic calculation of skin lesion areas between two consecutive measurements performed by the same investigator.

SECONDARY OUTCOMES:
Usability of the investigational software Clinicgram Euclides. | 1 day (at the end of the study)
  To evaluate the usability of the investigational software Clinicgram Euclides based on the completion of a usability questionnaire by each investigator who has used Clinicgram Euclides throughout the clinical investigation, and on the assessment of the time required to complete the calculation of the skin lesion area with each of the 3 methods (ruler measurement using Kundin method, investigational software Clinicgram Euclides, and digital planimetry using Adobe Photoshop).

CONTACTS AND LOCATIONS:
Overall Officials: María del Mar Martí Ejarque, Principal Investigator — Hospital University Sagrat Cor
Locations (1):
- Skilled Skin S.L., Barcelona, Spain